CLINICAL TRIAL: NCT05267821
Title: Targeted Reversal of Inflammation in Pediatric Sepsis-induced MODS (TRIPS)
Brief Title: Targeted Reversal of Inflammation in Pediatric Sepsis-induced MODS
Acronym: TRIPS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mark Hall, Chief, Division of Critical Care Medicine, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRIPS
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Sepsis-induced Multiple Organ Dysfunction Syndrome (MODS)
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Prospective, adaptively-randomized, double-blind, placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Anakinra 4 mg/kg/day (Active Comparator): IV Anakinra 4mg/kg/day x 7 days
  Interventions: Drug: Anakinra
- Anakinra 8 mg/kg/day (Active Comparator): IV Anakinra 8 mg/kg/day x 7 days
  Interventions: Drug: Anakinra
- Anakinra 12 mg/kg/day (Active Comparator): IV Anakinra 12 mg/kg/day x 7 days
  Interventions: Drug: Anakinra
- Anakinra 16 mg/kg/day (Active Comparator): IV Anakinra 16 mg/kg/day x 7 days
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): IV placebo x 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — See information in arm/group descriptions
  Arms: Anakinra 12 mg/kg/day; Anakinra 16 mg/kg/day; Anakinra 4 mg/kg/day; Anakinra 8 mg/kg/day
Drug: Placebo — See information in arm/group descriptions
  Arms: Placebo

SUMMARY:
The TRIPS study is a prospective, multi-center, double-blind, adaptively randomized, placebo-controlled clinical trial of the drug anakinra for reversal of moderate to severe hyperinflammation in children with sepsis-induced multiple organ dysfunction syndrome (MODS).

DETAILED DESCRIPTION:
The TRIPS study is a prospective, multi-center, double-blind, adaptively randomized, placebo-controlled clinical trial of the drug anakinra for reversal of moderate to severe hyperinflammation in children with sepsis-induced multiple organ dysfunction syndrome (MODS). Eligible subjects will undergo centralized immunophenotyping on day 2 of MODS. Subjects without immunoparalysis (a whole blood ex vivo LPS-induced TNF-alpha production capacity < 200 pg/ml) and a serum ferritin level of 500 - 2,000 ng/ml or a serum C-reactive protein (CRP) ≥ 4 mg/dl will be eligible for randomization, along with subjects with a serum ferritin level of 2,000 - 10,000 ng/ml regardless of their TNF-alpha response. Eligible subjects will receive intravenous (IV) anakinra at a dose of 4, 8, 12, or 16 mg/kg/day or placebo for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 weeks corrected gestational age to < 18 years; AND
* Admission to the PICU or CICU; AND
* Onset of ≥ 2 new organ dysfunctions within the last 3 calendar days (compared to pre-sepsis baseline) as measured by the modified Proulx criteria; AND
* Documented or suspected infection as the MODS inciting event.

Exclusion Criteria:

* Weight <3kg; OR
* Limitation of care order at the time of screening; OR
* Patients at high likelihood of progression to brain death in opinion of the clinical team; OR
* Moribund condition in which the patient is unlikely to survive the next 48 hours in opinion of the clinical team; OR
* Current or prior diagnosis of hemophagocytic lymphohistiocytosis or macrophage activation syndrome; OR
* Peripheral white blood cell count < 1,000 cells/mm3 as the result of myeloablative therapy OR receipt of myeloablative therapy within the previous 14 days; OR
* Known allergy to anakinra, or E. coli-derived products; OR
* Known pregnancy; OR
* Lactating females; OR
* Receipt of anakinra within the previous 28 days; OR
* Resolution of MODS by MODS Day 2; OR
* Previous enrollment in the TRIPS study.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative 28-day Pediatric Logistic Organ Dysfunction (PELOD-2) score | 28 days from randomization
  The cumulative Pediatric Logistic Organ Dysfunction (PELOD)-2 score over 28 days from randomization. The range of daily PELOD-2 scores is from 0 - 33, with higher scores representing worse organ function.

SECONDARY OUTCOMES:
3-month health-related quality of life | 3 months post-randomization
  The change in Pediatric Quality of Life inventory (PedsQL) score from baseline to 3-months post-randomization. The PedsQL score ranges from 0 - 100, with higher values indicating better quality of life.
3-month functional status | 3 months post-randomization
  The change in Functional Status Score (FSS) from baseline to 3-months post-randomization. The FSS score ranges from 6 - 30, with higher scores indicating worse functional status.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Benioff Children's Hospital - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, Davis, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Benioff Children's Hospital - Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Riley Children's Hospital, Indianapolis, Indiana
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mercy Children's Hospital, Kansas City, Missouri
  - Duke University, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] VanBuren JM, Hall M, Zuppa AF, Mourani PM, Carcillo J, Dean JM, Watt K, Holubkov R. The Design of Nested Adaptive Clinical Trials of Multiple Organ Dysfunction Syndrome Children in a Single Study. Pediatr Crit Care Med. 2023 Dec 1;24(12):e635-e646. doi: 10.1097/PCC.0000000000003332. Epub 2023 Jul 27. PMID 37498156